CLINICAL TRIAL: NCT03513393
Title: Influence of the Acidic Beverage Cola on the Absorption of the HCV Agent Velpatasvir in Healthy Volunteers Being Treated With the Proton Pump Inhibitor Omeprazole.
Brief Title: Influence of Cola on the Absorption of the HCV Agent Velpatasvir in Combination With PPI Omeprazole.
Acronym: COPA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: UMCN-AKF 17.02
Record Dates: First submitted 2018-04-18; First posted 2018-05-01 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2019-01

CONDITIONS: Hepatitis C; Swallowing Disorder
Keywords: velpatasvir; cola; omeprazole; proton pump inhibitors
MeSH Terms: conditions — Hepatitis C; Deglutition Disorders | interventions — velpatasvir; Omeprazole; Water

STUDY DESIGN:
Intervention Model Description: An open-label, 3-period, single-centre, phase-I, multi PPI dose, single velpatasvir dose trial in 12 healthy volunteers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- A: Epclusa + omeprazole + Coca Cola (test 1) (Experimental): Day 1 - 6 40mg omeprazole QD; on Day 5 a single-dose of SOF/VEL with 250 mL of Coca Cola Classic is administered (test 1).
  Interventions: Drug: velpatasvir
- B: Epclusa + omeprazole + water (test 2) (Experimental): Day 8 - 13: 40mg omeprazole QD; on Day 12 a single-dose of SOF/VEL is administered (test 2).
  Interventions: Drug: velpatasvir
- C: Epclusa + water (Reference) (Active Comparator): Day 15 - 21: no treatment with omeprazole; on Day 19 a single-dose of SOF/VEL is administered (reference).
  Interventions: Drug: velpatasvir

INTERVENTIONS:
Drug: velpatasvir — Test 1
  Other Names: Omeprazole; Coca Cola Classic 250ml
  Arms: A: Epclusa + omeprazole + Coca Cola (test 1)
Drug: velpatasvir — Test 2
  Other Names: Omeprazole; water 250ml
  Arms: B: Epclusa + omeprazole + water (test 2)
Drug: velpatasvir — Reference
  Arms: C: Epclusa + water (Reference)

SUMMARY:
Epclusa® is a pan-genotypic, once-daily tablet for the treatment of chronic hepatitis C virus (HCV) infection containing the NS5B- polymerase inhibitor sofosbuvir (SOF, nucleotide analogue) 400 mg and the NS5A inhibitor velpatasvir (VEL) 100 mg.

Velpatasvir has pH dependent absorption. At higher pH the solubility of velpatasvir decreases. It has been shown that in subjects treated with proton pump inhibitors (PPIs) such as omeprazole, the absorption of velpatasvir is reduced by 26-56%, depending on the dose of omeprazole, concomitant food intake, and timing/sequence of velpatasvir vs. omeprazole intake. As a result, concomitant intake of PPIs with velpatasvir is not recommended.

For a number of reasons, the prohibition of PPI use with velpatasvir is a clinically relevant problem. First, PPI use is highly frequent in the HCV-infected subject population with prevalences reported up to 40%. Second, PPIs are available as over-the-counter medications and thus can be used by subjects without informing their physician. Third, although HCV therapy is generally well tolerated, gastro-intestinal symptoms such as abdominal pain and nausea are frequently reported, which my lead to PPI use.

One solution of this problem could be the use of other acid-reducing agents such as H2-receptor antagonists or antacids. In general, they have a less pronounced effect on intragastric pH, and are considered less effective than PPIs by many patients and physicians.

A second solution would be the choice of another HCV agent or combination that is not dependent on low gastric pH for its absorption such as daclatasvir. Daclatasvir, however, is not a pan-genotypic HCV agent and may be less effective against GT 2 and 3 infections than velpatasvir. Second, not all subjects have access to daclatasvir, depending on health insurance company or region where they live.

A third solution, and the focus of this COPA study, is to add a glass of the acidic beverage cola at the time of velpatasvir administration in subjects concurrently treated with PPIs. This intervention has been shown to be effective for a number of drugs from other therapeutic classes who all have in common a reduced solubility (and thus reduced absorption) at higher intragastric pH, namely erlotinib, itraconazole, ketoconazole.

The advantages of this approach are: (1) only a temporary decrease in gastric pH at the time of cola intake; the rest of the day the PPI will have its therapeutic effect (2) cola is available worldwide (3) the administration of cola can be done irrespective to the timing of PPI use.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 and not older than 55 years at screening.
* Subject does not smoke more than 10 cigarettes, 2 cigars, or 2 pipes per day for at least 3 months prior to Day 1.
* Subject weighs at least 40 kg.
* Subject has a Quetelet Index (Body Mass Index) of 18 to 30 kg/m2, extremes included.
* Subject is able and willing to sign the Informed Consent Form prior to screening evaluations.
* Subject is in good age-appropriate health condition as established by medical history, physical examination, and electrocardiography, results of biochemistry, hematology and urinalysis testing within 4 weeks prior to Day 1. Results of biochemistry, hematology and urinalysis testing should be within the laboratory's reference ranges (see Appendix A). If laboratory results are not within the reference ranges, the subject is included on condition that the Investigator judges that the deviations are not clinically relevant. This should be clearly recorded.
* Subject has a normal blood pressure and pulse rate, according to the Investigator's judgment.

Exclusion Criteria:

* Creatinine clearance below 60 mL/min.
* Documented history of sensitivity/idiosyncrasy to medicinal products or excipients.
* Positive hepatitis B or C test
* Pregnant female (as confirmed by an hCG test performed less than 4 weeks before day 1) or breast-feeding female. Female subjects of childbearing potential without adequate contra-ception, e.g. hysterectomy, bilateral tubal ligation, (non-hormonal) intrauterine device, total abstinence, double barrier methods, or two years post-menopausal. They must agree to take precautions in order to prevent a pregnancy throughout the entire conduct of the study.
* Therapy with any drug (for two weeks preceding Day 1), except for acetaminophen (max 2 gram/day).
* Relevant history or presence of pulmonary disorders (especially COPD), cardiovascular disorders, neurological disorders (especially seizures and migraine), psychiatric disorders, gastro-intestinal disorders, renal and hepatic disorders (clinically relevant increased ALAT/ASAT or hyperbilirubinemia), hormonal disorders (especially diabetes mellitus), coagulation disorders.
* Relevant history or current condition that might interfere with drug absorption, distribution, metabolism or excretion.
* History of or current abuse of drugs, alcohol or solvents (positive drugs of abuse test).
* Inability to understand the nature and extent of the study and the procedures required.
* Participation in a drug study within 60 days prior to Day 1.
* Donation of blood within 60 days prior to Day 1.
* Febrile illness within 3 days before Day 1.
* Co-worker of Radboud university medical center.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Bioequivalence AUC0-inf | 21 days
  Determination of velpatasvir AUC0-inf by noncompartmental analysis.
  Descriptive statistics for the plasma concentrations of velpatasvir at each sampling time. Descriptive statistics for each PK parameter per treatment (geometric mean + CV%).
  Geometric Mean Ratios and 90% confidence intervals of pharmacokinetic parameters of A (Test 1) vs. C (Reference) and of B (Test 2) vs. C (Reference).
  AUC0-inf geometric mean ratios with a 90% Cl falling entirely within the range of 0.7 to 1.43 are considered bioequivalent.

SECONDARY OUTCOMES:
Safety and tolerability of Epclusa in healthy volunteers | 21 days
  To evaluate the safety and tolerability of SOFA/EL tablets in healthy volunteers.
  Adverse events after administration of SOFA/EL in the three interventions will be described and compared (including clinically relevant laboratory abnormalities).
Bioequivalence (Cmax) | 21 days
  Determination of velpatasvir Cmax by noncompartmental analysis.
Bioequivalence AUC0-48h | 21 days
  Determination of velpatasvir AUC0-48h by noncompartmental analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud university medical Center, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Result] van Seyen M, Colbers A, Abbink EJ, Drenth JPH, Burger DM. Concomitant Intake of Coca-Cola to Manage the Drug-Drug Interaction Between Velpatasvir and Omeprazole Studied in Healthy Volunteers. Clin Pharmacol Ther. 2019 Nov;106(5):1093-1098. doi: 10.1002/cpt.1569. Epub 2019 Aug 18. PMID 31313296
- See also: paper — https://pubmed.ncbi.nlm.nih.gov/31313296/